CLINICAL TRIAL: NCT01656265
Title: Phase I Study of ARQ 197 in Advanced Hepatocellular Carcinoma
Brief Title: Study of ARQ 197 in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARQ 197-008
Record Dates: First submitted 2012-07-20; First posted 2012-08-02 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Advanced Hepatocellular Carcinoma
MeSH Terms: interventions — ARQ 197

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ARQ 197 (Experimental)
  Interventions: Drug: ARQ 197

INTERVENTIONS:
Drug: ARQ 197 — Daily repeating dose of oral ARQ 197, twice a day just after meals. Dose of ARQ 197 will be escalated according to 3+3 rule.
  Other Names: Tivantinib

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of ARQ 197 in hepatocellular carcinoma (HCC) patients treated with daily oral ARQ 197, to determine the recommended dose of ARQ 197 in advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HCC patients who are resistant to, intolerable to, or rejecting a systemic sorafenib therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Child-Pugh classification A at the time of registration
* Adequate bone marrow, liver, and renal functions within 14 days prior to registration

Exclusion Criteria:

* Prior therapy with a c-Met inhibitor (including ARQ 197)
* Any systemic anti-tumor treatment or investigational agent within 2 weeks prior to registration. If the treatment/agent was antibody, within 4 weeks
* Local treatment for malignancy within 4 weeks prior to registration
* Major surgical procedure within 4 weeks prior to registration

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2012-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicity (DLT), as a measure of safety and tolerability | DLT observation period will be the first 28 days after the start of ARQ 197 treatment.
  Adverse Event collection and assessment will be done for all treated subjects to assess the safety, tolerability. The grading for the severity of the adverse events will be determined according to CTCAE ver 4.0.

SECONDARY OUTCOMES:
Profiles of Pharmacokinetics | Plasma sample correction at pre-dose 1, 2, 4, 6, 10, 12 and 24 hours on day 1; at pre-dose, 1, 2, 4, 6, 10, 12 hours on day 15; and at pre-dose on day 29.
  maximum concentration (Cmax), area under the curve (AUC), half-life (t1/2), apparent clearance (Cl/F), and apparent volume of distribution in the terminal elimination phase (Vz/F).
Antitumor effects according to RECIST 1.1. | Every 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Kashiwa, Chiba, Japan